CLINICAL TRIAL: NCT02916082
Title: Use of Cervical Length Previous to the Use of Prostaglandins as a Tool to Predict Vaginal Birth in Pregnancies With > 41 Weeks Gestation.
Brief Title: Cervical Length Pre-induction as a Tool to Predict Vaginal Birth
Status: Completed | Type: Observational
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Coordinator of Research, Saint Thomas Hospital, Panama
Other Study IDs: 2015-288V2
Record Dates: First submitted 2016-09-25; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Cervical Length Measurement; Pregnancy, Prolonged
Keywords: Cervical length; Prolonged pregnancy; Vaginal birth
MeSH Terms: conditions — Pregnancy, Prolonged

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prolonged pregnancy: Pregnancies with 41 weeks or more of gestation determined by a reliable last menstrual period or early fetal ultrasound.
  Interventions: Procedure: Cervical length measurement

INTERVENTIONS:
Procedure: Cervical length measurement — Vaginal ultrasound to measure cervical length previous to use of prostaglandins.

SUMMARY:
To evaluate the value of measuring cervical length as a predictor of vaginal birth after induction of labor with prostaglandins in pregnancies with 41 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

* 41 weeks or more of gestational age
* Cervical length measured by a FMF certified physician

Exclusion Criteria:

* Any condition that could interfere with a possible vaginal birth (previous cesarean section, hypertensive disorders of pregnancies).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnancies with a gestational age of 41 weeks or more.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Vaginal Birth | 72 hours
  Number of vaginal births obtained after a measure of cervical length below 2,5 cms.

SECONDARY OUTCOMES:
Induction to delivery time | 72 hours
  Time (hours) between the application of a prostaglandin and termination of pregnancy (vaginal or cesarean).

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Thomas H, Panama City, Provincia de Panamá, Panama